CLINICAL TRIAL: NCT03688893
Title: Efficacy of Laser Application in Dental Bleaching: A Randomized Clinical Trial
Brief Title: Efficacy of Laser Application in Dental Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Caaguazu (Other)
Responsible Party: Principal Investigator, Julieta María Méndez Romero, Doctor in Dental Surgery, Professor of Research Methodology, Universidad Nacional de Caaguazu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1219-0122
Record Dates: First submitted 2018-09-21; First posted 2018-09-28 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Tooth Discoloration
Keywords: Bleaching; Laser; CIELCH
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: The investigators conducted a Randomized controlled trial (RCT) to study the effect of LASER in dental bleaching in 24 patients in Paraguay in 2015.
Who Masked: Outcomes Assessor
Masking Description: It was single blind; as the evaluator did not know what intervention the patient was assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser Application (Experimental): 35% Hydrogen Peroxide (Whitening HP, FGM SC Brazil) 40 minutes divided in two phases of 20 minutes each one (5 minutes colocation, 10 minutes Laser Application and 5 minutes moving the product) from premolar to premolar in superior and inferior teeth. Experimental
  Interventions: Device: Laser Application for Dental Bleaching
- No Laser Application (No Intervention): 35% Hydrogen Peroxide (Whitening HP FGM SC Brazil), 40 minutes divided in two phases of 20 minutes each one (5 minutes colocation, 10 minutes waiting and 5 minutes moving the product) from premolar to premolar in superior and inferior teeth. No Laser Application No Intervention

INTERVENTIONS:
Device: Laser Application for Dental Bleaching — The Laser used was the Whitening Lase II (DCM EQUIPMENTS).
  Arms: Laser Application

SUMMARY:
Objective: To establish the efficacy of laser application with chemical treatment in dental bleaching compared to chemical treatment alone.

Methods: The investigators conducted a randomized controlled trial (RCT), single blind (evaluator), in 24 patients randomized to laser and chemical intervention (12) or chemical intervention aloe (12). The commercial products used were Whiteness Hp 35% Hydrogen Peroxide and the LASER of DCM Equipments. The trial outcome measures were obtained using the Vita EasyShade Spectrophotometer and the International CIELCh system. To stablish differences before vs. after treatments and between groups, the T test and chi2 tests were applied.

DETAILED DESCRIPTION:
New technologies continue to be launched in the field of dental esthetics, especially for whitening, and many products advertise their efficacy. One new approach is the use of LASER technology which has been purported to be the most powerful font light for bleaching Diverse studies by different designs find different efficacies for LASER whitening Randomized clinical trials (RCT) are needed for the most rigorous confirmation of efficacy. RCT are able to control for characteristics that can cause bias, including factors related to dental care such as diet and cleaning behavior after the bleaching procedure. The investigators therefore conducted an RCT to make a side by side comparison of a LASER whitening technique with chemical bleaching versus chemical bleaching without LASER.

Intervention: After the patient was informed and sign the consent; a dental prophylaxis was done. Three days later the bleaching procedure started following the same protocol regarding to the time and product used (35% Hydrogen Peroxide Whitening HP, 40 minutes divided in two phases of 20 minutes each one) from premolar to premolar in superior and inferior teeth. The difference was that one of the intervention groups used the Laser for ten minutes (starting at the minute 5) and the other did not.. The Laser used was the Whitening Lase II (DCM EQUIPMENTS).

The measure of the color was done to the superior canines by just one evaluator in three stages: before bleaching (baseline), 15 minutes after bleaching, and three days after. It was done with the Vita Easyshade Spectrophotometer.

The dental sensitivity also was asked at the three time points; however, as an exclusion criterion the level had to be 0 to be entered into the study.

All the patients received verbal and written instructions about eating and cleaning behavior. Cleaning materials for the three days after procedure were given.

As the clinical endpoint, the difference in color was calculated using the international accepted system CIELCh (11,18-19). The formula is ∆E* = [(∆L*)2 + (∆C*)2 + (∆h*)2] ½; were L is Luminosity, C is Chroma and h is Hue.

A verbal numeric scale was used to determine the dental sensitivity with values from 0 to 3. The evaluator used the water and air from the dental chair syringe. The patient reports 0 for no sensitivity; 1 for slight sensitivity, 2 for moderate sensitivity, and 3 for severe sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who wanted to bleach or whiten their teeth.

Exclusion Criteria:

* Patients who have a color less than A2 according to the Vita Scale
* Patients with dental sensitivity
* caries or restorations
* periodontal disease
* dental abfraction or attrition
* pregnant women, smokers
* patients with orthodontics
* nauseous reflects
* patients who did not wish to sign the consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09-05 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2015-09-25 (Actual)

PRIMARY OUTCOMES:
Dental Color Stage 1(Before Intervention) | through study completion, an average of 3 days
  The measure of the color was done to the superior canines by just one evaluator. It was done with the Vita Easyshade Spectrophotometer. To improve precision off the data, measures were taken 3 times in all superior canines studied. The Investigators used the values L, C,H.
Dental Color Stage 2 (30 minutes after dental bleaching) | through study completion, an average of 3 days
  The measure of the color was done to the superior canines by just one evaluator. It was done with the Vita Easyshade Spectrophotometer. To improve precision off the data, measures were taken 3 times in all superior canines studied. The Investigators used the values L, C,H.
Dental Color Stage 3 (3 days after dental bleaching) | through study completion, an average of 3 days
  The measure of the color was done to the superior canines by just one evaluator. It was done with the Vita Easyshade Spectrophotometer. To improve precision off the data, measures were taken 3 times in all superior canines studied. The Investigators used the values L, C,H.
Change in Color (Stage 3 - Stage 1) | through study completion, an average of 3 days
  The difference in color was calculated using the international accepted system CIELCh (11,18-19). The formula is ∆E* = [(∆L*)2 + (∆C*)2 + (∆h*)2] ½; were L is Luminosity, C is Chroma and h is Hue. The higher difference in color will show the better intervention.
Change in Color (Stage 2 - Stage 1) | through study completion, an average of 3 days
  The difference in color was calculated using the international accepted system CIELCh (11,18-19). The formula is ∆E* = [(∆L*)2 + (∆C*)2 + (∆h*)2] ½; were L is Luminosity, C is Chroma and h is Hue. The higher difference in color will show the better intervention.

SECONDARY OUTCOMES:
Immediate Dental Sensitivity | through study completion, an average of 3 days
  The dental sensitivity was asked 15 minutes after bleaching using a scale: None sensitivity, light sensitivity, moderate sensitivity, severe sensitivity. Less sensitivity is going to be better.
Mediate Dental Sensitivity | through study completion, an average of 3 days
  The dental sensitivity was asked 3 days after bleaching using a scale: None sensitivity, light sensitivity, moderate sensitivity, severe sensitivity. Less Sensitivity is going to be better.

CONTACTS AND LOCATIONS:
Overall Officials: Julieta M Méndez, DDs, Principal Investigator — Facultad de Odontología Universidad Nacional de Caaguazú; Ulises A Villasanti Torales, DDs, Mgst, Study Director — Facultad de Odontología Universidad Nacional de Caaguazú
Locations (1):
- Facultad de Odontología Universidad Nacional de Caaguazú, Coronel Oviedo, International, Paraguay

IPD SHARING:
Plan to Share IPD: Yes
By email
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From the time the protocol is available in clinicaltrials.gov and with no limit of time
Access Criteria: Researchers that want to know about the study and use the protocol

REFERENCES:
- [Background] González Rosino B. Estudio clínico comparativo entre dos dispositivos de luz para blanqueamientos en clínica. 2014; [citado 17 de julio 2015]. Disponible en: http://eprints.ucm.es/27417/
- [Background] Giannini M, Hirata R, Coelho AS, de Oliveira VAP, Chan DCN. Agentes Blanqueadores y Técnicas Utilizadas en Consultorio. ROBYD [Internet]. 2013 enero-abril;II(1). [citado 22 de julio 2015]. Disponible en: www.rodyb.com/agentes---blanqueadores---y---tecnicas---utilizadas---en--consultorio---27/
- [Background] Henry RK, Bauchmoyer SM, Moore W, Rashid RG. The effect of light on tooth whitening: a split-mouth design. Int J Dent Hyg. 2013 May;11(2):151-4. doi: 10.1111/j.1601-5037.2012.00568.x. Epub 2012 Jul 12. PMID 22783981
- [Background] Dostalova T, Jelinkova H, Housova D, Sulc J, Nemec M, Miyagi M, et al. Diode laser-activatedbleaching. BrazDent J. 2004;15(Special Issue):3-8. [citado 27 de marzo 2016]. Disponible en: http://blackstar.forp.usp.br/bdj/bdj15si/pdf/v15sia01.pdf
- [Background] Wetter NU, Walverde D, Kato IT, Eduardo Cde P. Bleaching efficacy of whitening agents activated by xenon lamp and 960-nm diode radiation. Photomed Laser Surg. 2004 Dec;22(6):489-93. doi: 10.1089/pho.2004.22.489. PMID 15684748
- [Background] Alomari Q, El Daraa E. A randomized clinical trial of in-office dental bleaching with or without light activation. J Contemp Dent Pract. 2010 Jan 1;11(1):E017-24. PMID 20098962